CLINICAL TRIAL: NCT03749798
Title: To Collect and Compare Data With an Intraoperative Wavefront Device (HeLeNa) to a Standard Wavefront Device: an Explorative Pilot Study
Brief Title: Comparing an Intraoperative vs. a Standard Wavefront Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HeLeNa
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract; Wavefront measurement
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative wavefront measurement (Experimental): Patients will be measured with an intraoperative wavefront device during cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Intraoperative wavefront measurements will be carried out during cataract surgery

SUMMARY:
Comparison of intraoperative measured wavefront data with pre- and post-operative wavefront data.

DETAILED DESCRIPTION:
Different technologies are in use for measuring wavefront aberrations, such as Hartmann-Shack wavefront aberrometry, Tscherning aberrometry, Laser Raytracing and automatic retinoscopy. While Hartmann-Shack wavefront aberrometry, the most widespread of these techniques, uses a lenslet array to record distortions of light bundles coming from a single source form the retina, Tscherning aberrometry uses a matrix of pinholes. Laser Ray Tracing in contrast measures the aberration of a laser beam at different locations. All three systems compare distorsions of the measured light beams with a perfect optical system to calculate the wavefront errors. Repeatability of wavefront devices was studied in young healthy subjects and different devices have been compared to each other. These results do not represent the typical cataract patient. Several factors, such as tear film instability and pupil size, have an influence on the measurements and these factors may change significantly with age.

Intraoperative measured data could help to get a better information about wavefront aberrations.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Able to understand the patient information
* Willing to follow the instructions and attend all follow-up visits
* Willing to sign informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases that are likely to reduce the refractive outcome, such as pseudoexfoliation syndrome, traumatic cataract, severe corneal scars
* Previous ocular surgeries on the study eye
* Patients who are not able to cooperate, with eccentric fixation or insufficient ability to fixate (tremor, nystagmus)
* Pregnant or lactating women (pregnancy testing will be performed preoperatively on women of reproductive age)

Ages: 21 Years to 105 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Wavefront aberration measurements | 12 months
  Measurements of wavefront aberrations using an Hartmann-Shack device will be compared at different time points (pre-, intra-, postoperative).

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided